CLINICAL TRIAL: NCT06544837
Title: Multi-national, Multi-center, Randomized Controlled Trial to Evaluate the Clinical Utility of Non-invasive Endometrial Receptivity Test (Ora) in Patients With Implantation Failure
Brief Title: Trial to Evaluate the Clinical Utility of Non-invasive Endometrial Receptivity Test (Ora) in Patients With Implantation Failure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Inti Labs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IntiLabs
Record Dates: First submitted 2024-08-05; First posted 2024-08-09 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-02

CONDITIONS: IVF; Window of Implantation; microRNA; Implantation; Non-invasive Testing; Endometrial Receptivity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Embryo implantation according to standard procedures
- ora Test Group (Experimental): Embryo implantation according to endometrial receptivity test (ora) recommendations
  Interventions: Diagnostic Test: Window of Implantation

INTERVENTIONS:
Diagnostic Test: Window of Implantation — Determine the subject's window of implantation through testing and adjust the embryo implantation time
  Arms: ora Test Group

SUMMARY:
The adjustment of the timing of embryo transfer based on the endometrial receptivity profile and transferring embryo(s) of good quality with normal chromosomes (diagnosed by Preimplantation Genetic Testing for Aneuploidy, PGT-A) are the two main causes to improve the success of assisted reproduction treatments (ART). Previously, endometrial receptivity analysis was performed on women undergoing IVF treatment through an invasive endometrial tissue biopsy. The aim of this study is to determine the clinical benefits of ORA, a novel non-invasive endometrial receptivity test that determines the optimal time for embryo transfer through a blood draw instead of an invasive endometrial tissue biopsy. It is expected to recruit 1000 couples whose embryos will be analyzed by PGT-A and/or who are going to evaluate their endometrium expression profile for endometrial receptivity. The patients will be randomized into two groups, (1) Control group : undergoing PGT-A only; (2) Study group : the undergoing both PGT-A and ORA. ART will be performed based on the results of PGT-A and/or ORA. Reproductive success, such as implantation rates (IR), pregnancy rates (PR), ongoing pregnancy rates (OGP) and live birth rates (LBR) will be tracked and compared.

Preliminary results demonstrate that both PGT-A and ORA can contribute to reproductive success, improving implantation rates in patients with implantation failure. Our hypothesis suggests that PGT-A and ORA could improve the performance of ART in infertile patients.

ELIGIBILITY:
Inclusion Criteria:

* Experienced implantation failure with euploid or low-level mosaic (< 30%) embryos in the past two years.
* Female age 28-45 years.
* Consent to undergo a simulated cycle for non-invasive optimal implantation window testing.
* Plan to undergo a frozen embryo transfer cycle.
* Have at least one euploid or low-level mosaic (< 30%) frozen blastocyst.

Exclusion Criteria:

* Presence of uterine cavity abnormalities that may affect implantation, such as polyps, fibroids ≧4 cm, or hydrosalpinx
* Presence of systemic diseases that may affect reproductive techniques (e.g., autoimmune diseases)
* Body mass index (BMI) over 30 kg/m²

Ages: 28 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 1000 (Estimated)
Dates: Start 2024-06-22 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 6 weeks after embryo transfer
  Rate of Participants with one or more intrauterine gestational sacs after 6 weeks of estimated gestational age.

SECONDARY OUTCOMES:
Ongoing pregnancy rate | 12 weeks after embryo transfer
  Rate of Participants with fetal heartbeat after 12 weeks of gestation.
Live birth rate | 20 weeks after embryo transfer
  Rate of Participants with live birth, defined as the delivery of a live infant with signs of life after 20 weeks of gestation.

CONTACTS AND LOCATIONS:
Locations (1):
- Hanoi Hospital, Hanoi, Vietnam

DOCUMENTS (1):
  • Study Protocol (2024-01-10): https://cdn.clinicaltrials.gov/large-docs/37/NCT06544837/Prot_000.pdf